CLINICAL TRIAL: NCT02956902
Title: A Smartphone Intervention With Telemedicine Support for Management of Post-traumatic Stress Disorder: A Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ontario Shores Centre for Mental Health Sciences (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-107IF
Record Dates: First submitted 2016-11-03; First posted 2016-11-07 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: PostTraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Waiting list control (No Intervention)
- Intervention (Experimental): Clinician-supported smartphone application intervention
  Interventions: Other: Clinician supported smartphone application intervention

INTERVENTIONS:
Other: Clinician supported smartphone application intervention
  Arms: Intervention

SUMMARY:
This study tests whether people receiving clinician support to use a mobile application on their smartphone can manage their post-traumatic stress disorder (PTSD) symptoms better than those who do not. Half of the participants will receive the clinician supported smartphone application intervention and the other half will remain on the waiting list.

ELIGIBILITY:
Inclusion Criteria:

* on the waiting list for the Ontario Shores traumatic stress clinic;
* score ≥ 31 on the PCL-5
* have access to a smartphone or tablet to which they are willing to download the app.

Exclusion Criteria:

* active suicidal ideation

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Change in PTSD symptom severity | 8 weeks
  Change in PTSD checklist (PCL-5) score

SECONDARY OUTCOMES:
Clinically significant change in PTSD symptom severity | 8 weeks
  Proportion of participants with a PCL-5 score less than 31
Change in Depression Severity | 8 week
  Change in patient health questionnaire 9 (PHQ-9) score
Average App Use per Week (Intervention group only) | 8 weeks
  Self-report app use will be collected by the clinician at each of sessions 2-4 by asking "on average, how many times did you use the app per day (or per week, if less than once per day). The clinician will also ask which of the four main functions were used and which symptom management tools were used most and were most helpful.
Goal Achievement (Intervention group only) | 8 weeks
  At each of sessions 1-3, the clinician will help the participant set goals, which will be documented. At each of sessions 2-4 the clinician will ask the participant to self-report goal achievement, which will be documented
Clinician Fidelity to Protocol | 8 weeks
  A fidelity checklist has been created for this protocol, which will be completed over the course of the intervention. The form will be updated upon completion of each clinician session.